CLINICAL TRIAL: NCT02026206
Title: Skin Adhesive Low-level Light Therapy for Primary Dysmenorrhea: A Double-blind Randomized Controlled Trial
Brief Title: Low-level Light Therapy for Primary Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pusan National University (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Associate Professor, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNUYH-03-2011-005
Record Dates: First submitted 2013-12-31; First posted 2014-01-01 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-02

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary Dysmenorrhea; Pain
MeSH Terms: conditions — Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LLLT group (Experimental): low-level light therapy (LLLT) was self-performed for 20 min/day over 5 days prior to the expected onset of menstruation during three menstrual cycles.
  Interventions: Device: low-level light therapy
- Placebo-controlled group (Placebo Comparator): Placebo low-level light therapy (LLLT) was self-performed for 20 min/day over 5 days prior to the expected onset of menstruation during three menstrual cycles. The placebo LLLT device was identical to the active device but did not radiate light as the hole was blocked.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: low-level light therapy — we used a skin-adhesive LLLT device called the Color DNA-WSF (Color Seven Co., Seoul, Korea) which consists of body for power supply and two microprocessor-controlled light-emitting diodes. We selected two acupuncture points, conception vessel 4 (CV4; Guanyuan) and CV6 (Qihai), for treating dysmenorrhea. The participants attached the skin-adhesive LLLT device probes to both acupuncture points according to treatment schedule.
  Other Names: Color DNA-WSF
  Arms: LLLT group
Device: Placebo — we used a placebo skin-adhesive LLLT device called the Color DNA-WSF (Color Seven Co., Seoul, Korea) which consists of body for power supply and two microprocessor-controlled light-emitting diodes. We selected two acupuncture points, conception vessel 4 (CV4; Guanyuan) and CV6 (Qihai), for treating dysmenorrhea. The participants attached the placebo skin-adhesive LLLT device probes to both acupuncture points according to treatment schedule.
  Arms: Placebo-controlled group

SUMMARY:
The purpose of this study was to evaluate the effectiveness of a self-therapeutic approach of skin adhesive low-level light therapy (LLLT) in females with primary dysmenorrhea (PD).

DETAILED DESCRIPTION:
Study design: This was a prospective, randomized, double-blind, placebo-controlled, multi-centered trial carried out at two university hospitals. This clinical trial was approved by the Korea Food and Drug Administration and the Institutional Review Boards of the two hospitals.

Study process:

All patients gave informed written consent after being informed of the details of the study. Participants were permitted to take analgesics when severe or difficult to control pain occurred. Participants were randomized into either the LLLT or placebo control groups at the third visit. All participants underwent demographic and history taking, a physical examination, an obstetrics and gynecology examination, ultrasound, and laboratory tests. All participants were educated on how to use the device by demonstration and a picture-guided user manual.

During the second visit, the participants conducted a self-evaluation of pain intensity and quality of life after the next menstruation started (pre-treatment score) using the VAS and EQ-5D questionnaire. The third visit occurred at least 5-7 days from the date of the next menstruation, and a clinical primary nurse described how to use the medical equipment and devices when they were at home. All subjects were to perform the LLLT 20 min/day for 5 days from the start of menstruation. Within 3 days after menstruation started the subjects self-assessed their pain using the VAS after treatment (first post-treatment score). Subjects carried out the self-treatment in the same way at home 5-7 days before the start of their next period and then visited the hospital for the fifth time to record their pain on the VAS (second post-treatment score). As before, self-therapy was performed 5-7 days before the next menstruation started. The sixth visit occurred within 1-3 days after menstruation began, just as before, and all subjects performed the self-evaluation (third post-treatment score) using the EQ-5D questionnaire and VAS for menstrual pain intensity.

Statistical analysis:

All data are summarized as means ± standard deviation or as numbers with proportions. A p < 0.05 was considered to indicate significance. We decided that the therapeutic effect would be a > 30% reduction in the VAS value after treatment. The statistical analysis was conducted using the VAS assessment score after the third treatment as the primary endpoint. We used an independent t-test to evaluate differences in each group between VAS pain scores measured after the third treatment and baseline values. The influence of variance in each group after pre-treatment, primary treatment, secondary treatment, and tertiary treatment were verified through repeated-measures analysis of variance (ANOVA). We analyzed the differences in the EQ-5D in each group using analysis of covariance (ANCOVA). Age was considered a covariate. Any differences between the groups for the use of painkillers were analyzed by Fisher's exact test. If there was any difference in the use of pain killers between groups, the influence of pain killer use was closely checked by ANCOVA. A per-protocol (PP) analysis was used in our clinical trial to assess efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of primary dysmenorrhea.
* a self-reported visual analog scale (VAS) for menstrual pain intensity over 7 on a scale of 0-10.

Exclusion Criteria:

* diagnosis of a serious medical or psychiatric illness, endometriosis or uterine fibroids, uterine adenomyosis, those taking oral contraceptives within the last 1 month, those who were pregnant or in whom the pregnancy test was positive were excluded.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Il Shin, Ph.D., Principal Investigator — Pusan National University Yangsan Hospital; Gi-Youn Hong, Ph.D., Principal Investigator — Wonkwang University Hospital
Locations (2):
- South Korea (2):
  - Wonkwang University Hospital, Iksan
  - Pusan National University Yangsan Hospital, Yangsan

REFERENCES:
- [Background] Shin YI, Kim NG, Park KJ, Kim DW, Hong GY, Shin BC. Skin adhesive low-level light therapy for dysmenorrhoea: a randomized, double-blind, placebo-controlled, pilot trial. Arch Gynecol Obstet. 2012 Oct;286(4):947-52. doi: 10.1007/s00404-012-2380-9. Epub 2012 May 31. PMID 22648444
- [Derived] Hong GY, Shin BC, Park SN, Gu YH, Kim NG, Park KJ, Kim SY, Shin YI. Randomized controlled trial of the efficacy and safety of self-adhesive low-level light therapy in women with primary dysmenorrhea. Int J Gynaecol Obstet. 2016 Apr;133(1):37-42. doi: 10.1016/j.ijgo.2015.08.004. Epub 2015 Dec 2. PMID 26797192

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LLLT Group | Placebo-controlled Group
Started | 44 | 44
Completed | 40 | 36
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LLLT Group | Placebo-controlled Group | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (3.6) | 25.3 (4.4) | 24.6 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 44 | 44 | 88
self-reported visual analog scale (VAS) for menstrual pain intensity [Mean (Standard Deviation); unit: units on a scale] — The primary outcome was menstrual pain intensity described using a 0-10 VAS scale.
  The higher values represent a worse outcome. All data collected by self-reported sheet.
  units on a scale | 8.30 (1.05) | 8.27 (0.92) | 8.28 (0.98)
quality of life as assessed by the EQ-5D [Mean (Standard Deviation); unit: units on a scale] — The secondary outcome measures were quality of life as assessed by the EQ-5D (minimun 0.00, maximum 1.00). The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The subscales combined to compute a total score according to EQ-5D equation formula. The higher values represent a better outcome.All data collected by self-reported sheet.
  units on a scale | 0.74 (0.20) | 0.74 (0.28) | 0.74 (0.24)

OUTCOME MEASURES:

1. Primary Outcome: Dysmenorrheal Pain Severity
Description: The primary outcome was menstrual pain intensity described using a 0-10 VAS scale (minimum 0, maximum 10). The higher values represent a worse outcome. All data collected by self-reported sheet. Before treatment, the participants conducted a self-evaluation of pain intensity after the next menstruation started (pre-treatment score) using the VAS. After self-therapy on 3 menstrual cycles, the participants conducted a self-evaluation of pain intensity after the next menstruation started (post-treatment score) using the VAS.
Time Frame: within 3 months after treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LLLT Group | Placebo-controlled Group
Number analyzed (Participants) | 40 | 36
units on a scale | 3.88 (2.09) | 6.31 (1.82)

2. Secondary Outcome: Quality of Life
Description: The secondary outcome measures were quality of life as assessed by the EQ-5D (minimun 0.00, maximum 1.00). The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The subscales combined to compute a total score according to EQ-5D equation formula. The higher values represent a better outcome.All data collected by self-reported sheet. Before treatment, the participants conducted a self-evaluation of pain intensity and quality of life after the next menstruation started (pre-treatment score) using the EQ-5D questionnaire. After self-therapy on 3 menstrual cycles, the participants conducted a self-evaluation of quality of life after the next menstruation started (post-treatment score) using the EQ-5D questionnaire.
Time Frame: within 3 months after treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LLLT Group | Placebo-controlled Group
Number analyzed (Participants) | 40 | 36
units on a scale | 0.91 (0.09) | 0.84 (0.14)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the clinical trial period (6 months)
Arm/Group | LLLT Group | Placebo-controlled Group
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 1/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LLLT Group (N=44) | Placebo-controlled Group (N=44)
Amenorrhea (Endocrine disorders) | 0 (0) | 1 (1) — For two months in placebo group after treatment with placebo, amenorrhea occurred in the next menstrual cycle. The subjects were to stop using placebo medical equipment, but amenorrhea has lasted for two months. menstruation began without treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No